CLINICAL TRIAL: NCT04639037
Title: Tight Postoperative Control of Mean Arterial Pressure Using a Closed-loop System for Norepinephrine Administration: A Randomized Controlled Trial in Patients Admitted to the Intensive Care Unit After a Major Surgery.
Brief Title: Control Mean Arterial Pressure in the Intensive Care Unit
Acronym: COMAP-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: University of California, Irvine (Other); University of California, Los Angeles (Other); Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP200709
Record Dates: First submitted 2020-11-05; First posted 2020-11-20 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Hypotension
Keywords: Intraoperative hypotension; intensive care unit; hemodynamic management
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Active comparator (manual adjustment of vasopressor infusion) and Experimental (automated management of vasopressor infusion)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual adjustment of vasopressor (Active Comparator): Fluid and vasopressor will be managed as standard practice guided by the EV1000 monitoring device (manually infusion of both fluid and vasopressors) Objective being to maintain MAP within a target MAP range of 80-90 mmHg (fluid will be optimized and stroke volume index will be maintained within normal values)
  Interventions: Device: Manual adjustment of vasopressor
- Automated adjustment of vasopressor (Experimental): Fluid will be managed using the EV1000 monitoring in order to optimize stroke volume index and vasopressor will be automatically deliver by a closed-loop system to maintain the MAP within the target range of 80-90 mmHg
  Interventions: Device: Automated adjustment of vasopressor

INTERVENTIONS:
Device: Automated adjustment of vasopressor — The objective of this randomized controlled superiority study is to demonstrate that, in patients admitted to intensive care after a major surgery, tight control of MAP using a closed-loop system for vasopressor administration will result in MAP being more often within a MAP range of 80-90 mmHg compared to the same management without this automated closed-loop system (nurse adjustment of vasopressor administration)
  Arms: Automated adjustment of vasopressor
Device: Manual adjustment of vasopressor — Fluid and vasopressor will be delivered as standard of care (manual adjustment of both fluid and vasopressor infusion rate by the nurse)
  Arms: Manual adjustment of vasopressor

SUMMARY:
The goal of this randomized controlled trial is to compare two different strategies of postoperative mean arterial pressure (MAP) management (manual versus automated) in patients who underwent a major surgery and admitted in the intensive care unit or post-anesthesia care unit for postoperative care. The investigators hypothesis is that the automated group will spend more time in a predetermined target MAP range of 80-90 mmHg compared to the manual group.

DETAILED DESCRIPTION:
Although the correction of hypotension during the perioperative period should be a key goal, approximately 40% of overall mortality is still closely linked to the presence of perioperative hypotension which is responsible for significant morbidity particularly in patients undergoing major surgery. Indeed, inadequate management of perioperative hypotension remains an undeniable risk factor for morbidity and mortality. However, management of perioperative mean arterial pressure (MAP) is still suboptimal today. Indeed, the analysis of our database demonstrates that, on average, patient spends only 50-60 % of the treatment time within the predetermined MAP target. In about 10% of the treatment time, the patient is under-treated (hypotension) and 30% of the time, the patient is over-treated (hypertension).

The correction of hypotension is achieved using vasopressor drugs (mainly norepinephrine infusion). In 2017 a study published in the JAMA shows that patients with tightly controlled arterial pressure have fewer organ dysfunctions than those with standard blood pressure management. However, maintaining MAP within a narrow range involves regular manual adjustments of norepinephrine infusion doses by intensive care unit nurses. When a hypotension occurs, there is usually two main possible treatments (fluid or vasopressors). In the operating room, for patients undergoing major surgery, we usually optimize fluid and vasopressor titration using an advanced hemodynamic monitoring device "EV1000 monitor" (Edwards Lifesciences, Irvine USA).This monitoring device can also be connected to a computer that controls a norepinephrine infusion pump in order to tightly adjust the infusion of norepinephrine to the target MAP predetermined by the clinician in charge of the patients. We have recently demonstrated that the use of such system resulted in less intraoperative time in hypotension compared to manual management. However, in the postoperative period, in patients admitted in the intensive care unit after a major surgery and requiring tight control of MAP, such demonstration is still lacking.

Therefore, the objective of this randomized controlled superiority study is to demonstrate that, in patients admitted to intensive care unit or post-anesthesia care unit after a major surgery, tight control of MAP using a closed-loop system for vasopressor administration will result in MAP being more often within a predetermined MAP range of 80-90 mmHg compared to the same management without this automated closed-loop system (nurse adjustment of vasopressor administration).

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (>18 years)
* Patients in the intensive care or post-anesthesia care unit after a major surgery and requiring norepinephrine infusion to maintain a MAP of 80-90 mmHg.
* Patients equipped with an advanced hemodynamic monitoring device as standard of care during the surgery.
* Patient with a social security number

Exclusion Criteria:

* Patients refusing to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Percentage of treatment time with a mean arterial pressure within 80-90 mmHg | at DAY 0
  Percentage of treatment time in target (defined as a mean arterial pressure within 80-90 mmHg)

SECONDARY OUTCOMES:
Percentage of treatment time in hypertension (MAP > 90 mmHg) | at DAY 0
  Percentage of treatment time in hypertension (defined as a MAP > 90 mmHg)
Percentage of treatment time in hypotension (MAP < 80 mmHg) | at DAY 0
  Percentage of treatment time in hypotension (defined as a MAP < 80 mmHg)
Percentage of treatment time in hypotension (MAP < 65 mmHg) | at DAY 0
  Percentage of treatment time in hypotension (defined as a MAP < 65 mmHg) which is the usual population target to correct
Volume of fluid during the treatment time | at DAY 0
  Volume of fluid during the treatment time
Amount of vasopressor used during the treatment time | at DAY 0
  total amount of vasopressor (norepinephrine) used during the treatment time to maintain MAP within 80-90 mmHg
Length of stay in the intensive care unit | up to 24 hours
  length of stay in the intensive care unit (discharge at the discretion of the clinician in charge of the patient and not involved in the study protocol)

OTHER OUTCOMES:
mean Stroke volume index during the treatment time | at DAY 0
  mean stroke volume index during the treatment time
mean Cardiax index during the treatment time | at DAY 0
  mean cardiac index during the treatment time

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Bicêtre Hospital, Le Kremlin-Bicêtre
  - Paul Brousse Hospital, Villejuif